CLINICAL TRIAL: NCT03295669
Title: Continuous Monitoring of Right Ventricular Function, Based on the Correlation Between the C-X Segment of the Central Venous Pressure Curve, and the Echocardiographic Evaluation of Right Ventricular Systolic Function
Acronym: CourbePVC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ELLOUZE 2016
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2017-09

CONDITIONS: Heart Surgery; Ultrasonography Right Ventricle Systolic Function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Close analysis of right ventricular function is still not done by all clinicians, even though it is indispensable; notably in cardiovascular ICUs.

Right ventricular dysfunction is responsible for increased morbidity and marks a turning point in the patient's prognosis.

It is difficult to analyse, and is principally assessed using echocardiography and by measuring the peak of the S' wave with pulsed Doppler and by measuring the tricuspid annular plane systolic excursion (TAPSE) in the TM mode. New studies have shown the interest of using 2D strain as a marker of systolic and diastolic function of the right ventricle. Finally, the use of 3D ultrasound seems to be more reliable than cardiac MRI for fine analysis of the right ventricle, even though it is rarely used in routine practice.

Study of the right ventricle using ultrasonography alone requires experienced and available operators for closely repeated evaluations making it possible to detect right ventricle dysfunction quickly.

US monitoring of left and right heart function is done systematically and repeatedly during post-operative care following heart surgery. This US evaluation could be optimized by finding a way to monitor the right ventricle continuously.

From a physiological point of view, we know about the tight relationship between the aspect of the central venous pressure curve and more precisely the C-X segment (tricuspid bulging into the atrium and start of contraction of the right ventricle) and right ventricular function. We wish to analyse this segment, combined with a US evaluation, and to look for a possible correlation so as to allow continuous, easy-to-interpret monitoring of right ventricular systolic function.

This will be facilitated by the systematic presence of a central venous catheter in every patient undergoing heart surgery, thus allowing central venous pressure to be monitored.

To this end, we wish to collect different data from patients in the cardiovascular ICU, especially the central venous pressure curve, the ventilatory pressure curve and settings of the respirator, and to carry out an echography evaluation of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the cardiovascular ICU
* Patients with spontaneous breathing
* With a central venous catheter placed in the internal jugular vein and for whom the central venous pressure curve is exploitable
* With a US window allowing a 4-chamber view making it possible to calculate the right ventricle ejection fraction (Peak of the S' wave, of the TAPSE, Strain of the right ventricle)

Exclusion Criteria:

* Non-echogenic patients or those without an exploitable US window
* Patients without a central venous catheter in the internal jugular vein
* Patients with an unexploitable central venous pressure curve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a cardiovascular ICU following heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Measure the peak of the S' wave | At baseline
Measure the tricuspid annular plane systolic excursion (TAPSE) | At baseline
Calculate strain in the right ventricle | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France